CLINICAL TRIAL: NCT02842060
Title: Development of a Tailored HIV Prevention Intervention for Young Men
Acronym: myDEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Jose Bauermeister, Presidential Associate Professor of Nursing, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34MH101997 (NIH)
Record Dates: First submitted 2016-07-16; First posted 2016-07-22 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: HIV Infections
Keywords: Prevention & Control; Young Adult; Internet
MeSH Terms: conditions — HIV Infections | interventions — N-nitroso-1,2,3,6-tetrahydropyridine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- myDEx Intervention (Experimental): The proposed intervention will consist of a 6-session web-based program. Cognizant of challenges maintaining users' attention in a web application and to facilitate delivery through a smartphone, the investigators will design each session to be no more than 20 minutes in length. In the course of these 6 sessions, YMSM will have a total of 120 minutes of intervention exposure. Across sessions, the investigators will emphasize the importance of sexual decision-making across different partner types, help YMSM consider what type of relationship(s) they want, and align these relationship desires with safer sex practices.
  Interventions: Behavioral: myDEx
- Non-tailored HIV Prevention (Active Comparator): The investigators will create a 6-session web-based attention-control comparison to match myDEx in time and attention yet have non-tailored and non-interactive content (NTHP). NTHP will include HIV/STI information currently available on sex education websites.
  Interventions: Behavioral: NTHP

INTERVENTIONS:
Behavioral: myDEx — myDEx will consist of a 6-session online program. Cognizant of challenges maintaining users' attention in a web application and to facilitate delivery through a smartphone, the investigators will design each session to be no more than 20 minutes in length. In the course of these 6 sessions, participants will have a total of 120 minutes of intervention exposure. Across sessions, the investigators will emphasize the importance of sexual decision-making across different partner types, help men consider what type of relationship(s) they want, and align these relationship desires with safer sex practices.
  Arms: myDEx Intervention
Behavioral: NTHP — The investigators will create a 6-session attention-control comparison to match the intervention in time and attention yet have non-tailored and non-interactive content (NTHP). NTHP will include HIV/STI information currently available on sex education websites. The attention-control condition allows the investigators to avoid confounding due to content and ensures that all participants receive some HIV prevention content given their high vulnerability to HIV. Further, this comparison will help critically examine the extent to which tailoring increases the acceptability to the program, above and beyond having a non-tailored, non-interactive intervention.
  Arms: Non-tailored HIV Prevention

SUMMARY:
This study uses an interactive design and development process to develop tailored messages that align YMSM's relationship experiences and desires with HIV prevention strategies. The study includes a tailored online prevention, intervention, as well as an attention control non--tailored HIV prevention (NTHP) comparison intervention. The pilot RCT will compare the intervention (N=120) to NTHP (N=60) to assess intervention feasibility and acceptability, and gather preliminary behavioral data to inform a subsequent application. Follow-up assessments will be collected at thirty (30), sixty (60), and ninety (90) days post-intervention.

DETAILED DESCRIPTION:
A resurgence of new HIV cases among young men who have sex with men (YMSM; ages 18--24) has underscored the importance of developing culturally- and developmentally- informed HIV programs for YMSM. The investigators are developing and pilot testing a tailored, web- based intervention called myDEx that focuses on delivering HIV prevention messages based on single YMSM's relationship expectations and partner--seeking behaviors. To maximize intervention appeal and appropriateness, the investigators have convened a youth advisory board (YAB) to provide insight and feedback during the 3--stage intervention development process. Using an iterative design and development process, they have developed tailored messages that align YMSM's relationship experiences and desires with HIV prevention strategies. The investigators designed and developed the myDEx tailored online prevention intervention, as well as an attention- control non--tailored HIV/AIDS prevention (NTHP) comparison intervention. After developing both interventions, the investigators used usability testing procedures to collect preliminary data from 16 YMSM on the proposed intervention's design and acceptability. Recommended changes were added to the intervention prior to launching a small pilot randomized controlled trial (RCT). The pilot RCT will compare myDEx (N=120) to NTHP (N=60) to assess intervention feasibility and acceptability, and gather preliminary behavioral data to inform a subsequent application. Assessments will be collected at 30, 60, and 90 days follow--up.

Specific Aims include:

1. To develop a tailored (myDEx) and non-tailored (NTHP) HIV prevention intervention focused on addressing HIV risk behaviors among single YMSM;
2. To collect preliminary data on the feasibility, acceptability, and intervention content of the myDEx (N=16) in preparation for a small pilot RCT; and,
3. To implement a small pilot RCT of the refined myDEx (N=120) as compared to the NTHP (N=60) intervention, in order to evaluate its feasibility and acceptability and gather preliminary efficacy results in reducing sexual risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Cis-gender male
* Self-report as being single
* Self report as HIV-negative at baseline
* Speak and read English
* Report unprotected anal intercourse with a male partner in prior six (6) months
* Have access to computer or smartphone device

Exclusion Criteria:

* Transgender identity
* HIV positive diagnosis
* Not residing in the United States
* Does not engage in male-to-male sexual behavior

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Bauermeister, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will assure the timely release and sharing of data two years after the publication of the main trial findings from the final dataset. Study variables will be available; however, the investigators will protect the rights and privacy of human subjects by redacting all identifiers from the dataset. The de-identified data from this project will be available through individual requests directed to the Principal Investigator.

REFERENCES:
- [Derived] Choi SK, Golinkoff J, Michna M, Connochie D, Bauermeister J. Correlates of Engagement Within an Online HIV Prevention Intervention for Single Young Men Who Have Sex With Men: Randomized Controlled Trial. JMIR Public Health Surveill. 2022 Jun 27;8(6):e33867. doi: 10.2196/33867. PMID 35759333
- [Derived] Connochie D, Tingler RC, Bauermeister JA. Young men who have sex with men's awareness, acceptability, and willingness to participate in HIV vaccine trials: Results from a nationwide online pilot study. Vaccine. 2019 Oct 8;37(43):6494-6499. doi: 10.1016/j.vaccine.2019.08.076. Epub 2019 Sep 13. PMID 31522806
- [Derived] Bauermeister JA, Tingler RC, Demers M, Harper GW. Development of a Tailored HIV Prevention Intervention for Single Young Men Who Have Sex With Men Who Meet Partners Online: Protocol for the myDEx Project. JMIR Res Protoc. 2017 Jul 19;6(7):e141. doi: 10.2196/resprot.7965. PMID 28724513

RESULTS

PARTICIPANT FLOW:
Groups:
- myDEx Intervention: The proposed intervention will consist of a 6-session web-based program. Across sessions, the investigators will emphasize the importance of sexual decision-making across different partner types, help YMSM consider what type of relationship(s) they want, and align these relationship desires with safer sex practices.
  myDEx: myDEx will consist of a 6-session online program. Cognizant of challenges maintaining users' attention in a web application and to facilitate delivery through a smartphone, the investigators will design each session to be no more than 20 minutes in length. In the course of these 6 sessions, participants will have a total of 120 minutes of intervention exposure. Across sessions, the investigators will emphasize the importance of sexual decision-making across different partner types, help men consider what type of relationship(s) they want, and align these relationship desires with safer sex practices.
Period: Overall Study
Arm/Group | myDEx Intervention | Non-tailored HIV Prevention
Started | 120 | 60
Completed | 120 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | myDEx Intervention | Non-tailored HIV Prevention | Total
Number analyzed (Participants) | 120 | 60 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.57 (1.81) | 21.87 (1.78) | 21.67 (1.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 120 | 60 | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 19 | 54
  Not Hispanic or Latino | 85 | 41 | 126
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 7 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 6 | 18
  White | 81 | 40 | 121
  More than one race | 20 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 120 | 60 | 180
Current PrEP Use [Count of Participants; unit: Participants] | 17 | 8 | 25
Receptive Anal Sex (past 30 days) [Count of Participants; unit: Participants] | 70 | 40 | 110
Alcohol use before/during sex (past 30 days) [Count of Participants; unit: Participants] | 43 | 27 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change in Number of Risky Sexual Partnerships
Description: The investigators estimated the change in the total number of participants who reported engaging in condomless anal intercourse from baseline to 90-day follow-up.
Time Frame: Count of participants from baseline to 90-day follow-up reported
Measure: Count of Participants; unit: Participants
Arm/Group | myDEx Intervention | Non-tailored HIV Prevention
Number analyzed (Participants) | 120 | 60
Participants
  Engaged in Condomless Receptive Anal Sex | 32 | 24
  No Condomless Receptive Anal Sex | 88 | 36

2. Primary Outcome: Number of Participants With Change in HIV Testing Behavior
Description: The investigators estimated the number of participants who reported testing for HIV from baseline to 90-day follow-up.
Time Frame: Count of participants from baseline to 90-day follow-up reported
Measure: Count of Participants; unit: Participants
Arm/Group | myDEx Intervention | Non-tailored HIV Prevention
Number analyzed (Participants) | 120 | 60
Participants | 56 | 29

3. Secondary Outcome: Change in Self-efficacy Motivations to Engage in HIV Prevention Behaviors
Description: The investigators will measure the change in safer sex self-efficacy over time using the HIV Risk Behavior Self-Efficacy Scale by Fisher, Fisher, Misovich, Kimble & Malloy (1996). The scale is measured on a 4-point scale (range 1-4), where higher scores mean less self-efficacy to negotiate safer sex with partners met online.
Time Frame: Baseline to 90-day follow-up period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | myDEx Intervention | Non-tailored HIV Prevention
Number analyzed (Participants) | 95 | 51
score on a scale | 1.93 (.56) | 1.99 (.49)

4. Secondary Outcome: Changes in Psychological Well-being
Description: The investigators will measure symptoms of depression and anxiety using the Brief Symptom Inventory by Derogatis & Spencer (1982). Higher mean scores (scale 1-4) indicate greater symptoms of psychological distress.
Time Frame: Baseline to 90-day follow-up period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | myDEx Intervention | Non-tailored HIV Prevention
Number analyzed (Participants) | 94 | 51
score on a scale | 1.84 (.58) | 1.93 (.66)

ADVERSE EVENTS:
Time Frame: 3-months
Description: The study was minimal risk. No participant reported any adverse event information to the study team.
Arm/Group | myDEx Intervention | Non-tailored HIV Prevention
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/60
Other Adverse Events (participants affected / at risk) | 0/120 | 0/60

LIMITATIONS AND CAVEATS:
We did not include biological confirmation of HIV/STI status through serologic tests, as this pilot trial did not seek to detect statistical differences in outcomes. HIV testing will be included in a full-scale efficacy trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT02842060/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT02842060/ICF_001.pdf